CLINICAL TRIAL: NCT05992350
Title: Garmin PACT (Physical Activity Tracking)
Brief Title: Garmin PACT (Physical Activity Tracking in Type 1 Diabetes Using Garmin Vivosmart)
Status: Terminated | Type: Observational
Why Stopped: Staffing shortages
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00002582
Record Dates: First submitted 2023-05-23; First posted 2023-08-15 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Garmin physical activity tracker — The Garmin physical activity tracker is worn like a watch on the user. The tracker assesses several physical states, indicates when the body is at optimal time for activity or when the body needs to rest. The tracker also monitors stress levels and prompts relaxation when appropriate. The tracker sets goals with participants based on previously completed activity. The tracker alerts participants after a period of inactivity, encourages regular movement throughout the day, and decreases the amount of time spent sedentary.

SUMMARY:
The goal of this observational study is to test the Garmin Vivosmart in children and youth (8-21) with Type 1 Diabetes (T1D) and their parents. The main questions it aims to answer are:

* Does the Garmin Vivosmart increase physical activity (PA)?
* Does the Garmin Vivosmart improve T1D status

Participants will:

* Wear the Garmin Vivosmart (4 or higher) for a year
* Complete surveys at the beginning, middle and end of participation asking about your T1D, T1D management, and PA
* Parents of children will also complete similar surveys about T1D

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 8-21 years of age and/or parent of participant aged 8-17 years of age
* Participants diagnosed with T1D greater than 6 months ago
* Participants must be patients at the Children's Mercy Kansas City network

Exclusion Criteria:

* Participants who do not meet age criteria above
* Participants who do not have T1D
* Participants who are unwilling to wear the device for at least 6 months

Ages: 8 Years to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Youth (8-21 YO) diagnosed with T1D and parents of youth (8-17 YO)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clements, MD, Principal Investigator — Children's Mercy
Locations (1):
- Children's Mercy, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cescon M, Choudhary D, Pinsker JE, Dadlani V, Church MM, Kudva YC, Doyle Iii FJ, Dassau E. Activity detection and classification from wristband accelerometer data collected on people with type 1 diabetes in free-living conditions. Comput Biol Med. 2021 Aug;135:104633. doi: 10.1016/j.compbiomed.2021.104633. Epub 2021 Jul 12. PMID 34346318
- [Background] Grimes A, Lightner JS, Eighmy K, Steel C, Shook RP, Carlson J. Decreased Physical Activity Among Youth Resulting From COVID-19 Pandemic-Related School Closures: Natural Experimental Study. JMIR Form Res. 2022 Apr 15;6(4):e35854. doi: 10.2196/35854. PMID 35297778
- [Background] Jaggers JR, McKay T, King KM, Thrasher BJ, Wintergerst KA. Integration of Consumer-Based Activity Monitors into Clinical Practice for Children with Type 1 Diabetes: A Feasibility Study. Int J Environ Res Public Health. 2021 Oct 10;18(20):10611. doi: 10.3390/ijerph182010611. PMID 34682355
- [Background] Ozaslan B, Patek SD, Breton MD. Impact of Daily Physical Activity as Measured by Commonly Available Wearables on Mealtime Glucose Control in Type 1 Diabetes. Diabetes Technol Ther. 2020 Oct;22(10):742-748. doi: 10.1089/dia.2019.0517. PMID 32105515

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only parent data was collected for Secondary Outcomes 16, 18, and 21. Parents only completed the Hypoglycemic Fear Scale II for Parents (HFS-P).
Groups:
- Primary Analysis Arm: Youth (8-21 YO) diagnosed with T1D.
- Parent Arm: Parents of youth (8-18YO) diagnosed with T1D.
Period: Overall Study
Arm/Group | Primary Analysis Arm | Parent Arm
Started | 24 | 21
Completed | 3 | 0
Not Completed | 21 | 21

BASELINE CHARACTERISTICS:
Population: Only parent data was collected for Secondary Outcomes 16, 18, and 21. Parents only completed the Hypoglycemic Fear Scale II for Parents (HFS-P).
Groups:
- Parent Arm: Parents of youth (8-18 YO) diagnosed with T1D
- Total: Total of all reporting groups
Arm/Group | Primary Analysis Arm | Parent Arm | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants] — Population: Only parent data was collected for Secondary Outcomes 16, 18, and 21. Parents only completed the Hypoglycemic Fear Scale II for Parents (HFS-P).
  Participants
    number analyzed (Participants) | 24 | 0 | 24
    <=18 years | 3 |  | 3
    Between 18 and 65 years | 21 |  | 21
    >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only parent data was collected for Secondary Outcomes 16, 18, and 21. Parents only completed the Hypoglycemic Fear Scale II for Parents (HFS-P).
  Participants
    number analyzed (Participants) | 24 | 0 | 24
    Female | 10 |  | 10
    Male | 14 |  | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only parent data was collected for Secondary Outcomes 16, 18, and 21. Parents only completed the Hypoglycemic Fear Scale II for Parents (HFS-P).
  Participants
    number analyzed (Participants) | 24 | 0 | 24
    Hispanic or Latino | 3 |  | 3
    Not Hispanic or Latino | 17 |  | 17
    Unknown or Not Reported | 4 |  | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only parent data was collected for Secondary Outcomes 16, 18, and 21. Parents only completed the Hypoglycemic Fear Scale II for Parents (HFS-P).
  Participants
    number analyzed (Participants) | 24 | 0 | 24
    American Indian or Alaska Native | 0 |  | 0
    Asian | 0 |  | 0
    Native Hawaiian or Other Pacific Islander | 0 |  | 0
    Black or African American | 4 |  | 4
    White | 19 |  | 19
    More than one race | 1 |  | 1
    Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Moderate to Vigorous Physical Activity (MVPA) Amount
Description: Minutes per Day of MVPA
Time Frame: Up to 365 days +- 30 days
Population: Study terminated before analysis took place, due to slow enrollment and unexpected termination the little data collected could not be analyzed. There is no future plan to analyze the data.
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

2. Primary Outcome: Diabetic Ketoacidosis (DKA) Admission
Description: Rate of hospitalization for diabetic ketoacidosis
Time Frame: 90 days +- 30 days
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

3. Primary Outcome: Diabetic Ketoacidosis (DKA) Admission
Description: Rate of hospitalization for diabetic ketoacidosis
Time Frame: 180 days +- 30 days
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

4. Primary Outcome: Diabetic Ketoacidosis (DKA) Admission
Description: Rate of hospitalization for diabetic ketoacidosis
Time Frame: 365 +-30 days
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

5. Primary Outcome: Change in Time in Range
Description: Time where blood glucose is in an appropriate range (and other glucose measurements)
Time Frame: Over 90, 180, and 365 +- 30 days
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

6. Primary Outcome: Predicted Change
Description: machine learning models to predict change in HbA1c, DKA admissions, and change in Time in Range
Time Frame: 90 +- 30 days
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

7. Primary Outcome: Predicted Change
Description: machine learning models to predict change in HbA1c, DKA admissions, and change in Time in Range
Time Frame: 180 +- 30 days
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

8. Primary Outcome: Predicted Change
Description: machine learning models to predict change in HbA1c, DKA admissions, and change in Time in Range
Time Frame: 365 +- 30 days
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

9. Primary Outcome: Minutes of Sleep Per Day
Description: Minutes of Sleep per Day
Time Frame: Up to 365 days +- 30 days
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

10. Secondary Outcome: Self Reported Physical Activity
Description: Self-reported physical activity via the International Physical Activity Questionnaire Short Form (IPAQ-SF), no min or max, recording the amount of time spent in MVPA in the past week, higher amounts are better.
Time Frame: 0 months
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

11. Secondary Outcome: Self Reported Physical Activity
Description: Self-reported physical activity via the International Physical Activity Questionnaire Short Form (IPAQ- SF), no min or max, recording the amount of time spent in MVPA in the past week, higher amounts are better.
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

12. Secondary Outcome: Self Reported Physical Activity
Description: Self-reported physical activity via the International Physical Activity Questionnaire Short Form (IPAQ-SF), no min or max, recording the amount of time spent in MVPA in the past week higher amounts are better.
Time Frame: 12 months
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

13. Secondary Outcome: Self Reported T1D Management
Description: Hypoglycemic Fear Scale (HFS-II) min 0 max 132, higher scores are a worse outcome
Time Frame: 0 months
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

14. Secondary Outcome: Self Reported T1D Management
Description: Hypoglycemic Fear Scale (HFS-II) min 0 max 132, higher scores are a worse outcome
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

15. Secondary Outcome: Self Reported T1D Management
Description: Hypoglycemic Fear Scale (HFS-II) min 0 max 132, higher scores are a worse outcome
Time Frame: 12 months
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

16. Secondary Outcome: Self Reported T1D Management
Description: Hypoglycemic Fear Scale II for Parents (HFS-P) min 0 max 143, higher scores are a worse outcome
Time Frame: 0 months
Population: as for outcome 1
Groups:
- Primary Analysis Arm: Parents of youth (8-21 YO) diagnosed with T1D
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

17. Secondary Outcome: Self Reported T1D Management
Description: Hypoglycemic Fear Scale II for Parents (HFS-P) min 0 max 143, higher scores are a worse outcome
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

18. Secondary Outcome: Self Reported T1D Management
Description: Hypoglycemic Fear Scale II for Parents (HFS-P) min 0 max 143, higher scores are a worse outcome
Time Frame: 12 months
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

19. Secondary Outcome: Change in Self Reported Physical Activity Levels
Description: Change in self reported physical activity levels via self-report with the IPAQ survey no min or max, recording the amount of time spent in MVPA in the past week, higher amounts are better.
Time Frame: Between 0, 6, and 12 months
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

20. Secondary Outcome: Change in How Participants Feel About Episodes of Hypoglycemia
Description: Change in how participants feel about episodes of hypoglycemia measured via the Hypoglycemic Fear Scale II (HFS-II) min 0 max 132, higher scores are a worse outcome
Time Frame: Between 0, 6, and 12 months
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

21. Secondary Outcome: Change in How Parents Feel About Episodes of Hypoglycemia in Their Children
Description: Change in how parents feel about episodes of hypoglycemia in their children wearing the Garmin physical activity tracker via the Hypoglycemic Fear Scale II for Parents (HFS-P) min 0 max 143, higher scores are a worse outcome
Time Frame: Between 0, 6, and 12 months
Population: as for outcome 1
Arm/Group | Primary Analysis Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Only adverse events were monitored for youth as parents only completed Hypoglycemic Fear Scale II for Parents (HFS-P) for the study.
Arm/Group | Primary Analysis Arm
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 3/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Analysis Arm (N=24)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT05992350/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT05992350/ICF_001.pdf